CLINICAL TRIAL: NCT02484027
Title: Effect of Rosuvastatin on Prognosis of Clinical Response in Acute Ischemic Stroke Patients
Brief Title: Effect of Rosuvastatin on Prognosis of Clinical Response in Acute Ischemic Stroke Patients(REPAIRS)
Acronym: REPAIRS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Collaborators: Taicang No.1 People's hospital (Unknown); AstraZeneca (Industry); National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Chun-Feng Liu, Associate Dean, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10580
Record Dates: First submitted 2015-06-17; First posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Infarction, Anterior Cerebral Artery
Keywords: acute ischemic stroke; mRS; rosuvastatin
MeSH Terms: conditions — Infarction, Anterior Cerebral Artery; Ischemic Stroke | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- statin-therapy (Experimental): Rosuvastatin orally at a dose of 20mg daily is assigned to patients immediately for the first 3 days of hospitalization. From the fourth day onward, rosuvastatin 10 mg daily will be administered for 1 year.
  Interventions: Drug: Rosuvastatin
- non-statin-therapy (Sham Comparator): No statins is assigned to patients for the first 3 days of hospitalization. From the fourth day onward, rosuvastatin 10 mg daily will be administered for 1 year.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Patients will be randomly assigned to receive 2 different therapies for the first 3 days of hospitalization: no statins (non-statin-therapy group) or to immediately receive rosuvastatin orally at a dose of 20mg daily (statin-therapy group). From the fourth day onward, rosuvastatin 10 mg daily will be administered in all patients for 1 year

SUMMARY:
This study is randomized, open-lable, parallel-group and comparator-controlled. 456 consecutive patients with acute ischemic stroke admitted within the first 72 hours after onset of symptoms will be studied. Those patients who will be randomly assigned to receive 2 different treatment for the first 3 days of hospitalization(non-statin-therapy group) or to immediately receive rosuvastatin orally at a dose of 20mg daily (statin-therapy group). From the fourth day onward, rosuvastatin 10 mg daily will be administered in all patients. The total trial will be continued 12 months.

mRS will be investigated at baseline, 3rd month, 12th month ;MMSE and Montreal tests will be investigated at baseline and 12th month. Laboratory data including serum lipids, Fg and hs-CRP.Among these, serum lipids will be tested at baseline, 8th day, 3rd month, 6th month,and 12th month; hs-CRP will be tested at baseline and 8th day, 3rd month; Fg will be tested at baseline, 8th day, 3rd month. Safety will be also assessed by adverse event reports and clinical laboratory data including CK-MB, renal and hepatic function at 3rd month, 6th month,12th month.

DETAILED DESCRIPTION:
This study is randomized, open-lable, parallel-group and comparator-controlled.456 consecutive patients with anterior circulation ischemic stroke within 72h from 2 participating hospitals are enrolled into the study. Those patients who will be randomly assigned to receive 2 different treatments for the first 3 days of hospitalization(non-statin-therapy group) or to immediately receive rosuvastatin orally at a dose of 20mg daily (statin-therapy group). From the fourth day onward, rosuvastatin 10 mg daily will be administered in all patients. The total trial will be continued 12 months.Subject eligibility will be established before treatment randomization. A random number table will be generated using a computerized procedure and subjects will be randomized strictly sequentially as they are eligible for randomization. The randomization procedure will be done like this. The random number will be divided by 2. And if the remainder is 1, the subject will be assigned to intensive rosuvastatin group. Correspondingly, if the remainder is 0, the subject will be assigned to the non-rosuvastatin group. Subjects will be randomized on a 1:1 schedule.

According to the previous post hoc analysis and SPARCL analysis results, the mRS event rate (mRS>2) at 90 days among statin-naïve patients before admission is 42% without statin treatment in the first 3 days of admission versus 28% with statin immediately used since admission. Previous studies showed there is benefit with statin treatment in the earlier period of acute ischemic stroke, so the data from SPARCL reserved conservatively because the patients within 6 months of stroke onset were enrolled. It is based on these reported event rates, a sample size of 182 patients per group will have 80% power to detect a rate difference of 14%, assuming a null rate difference of zero and using Pearson's chi-squared test with a two-sided significance level of 0.05. With an estimated 20% rate of dropping out from the study, a total of 456 patients will have to be randomized (228 in each group) for this study.

Medical histories were obtained from all subjects before enrollment. Patients are followed by 1 year. mRS will be investigated at baseline, 3rd month, 12th month ;MMSE and Montreal tests will be investigated at baseline and 12th month. Laboratory data include serum lipids, Fg and hs-CRP.Among these, serum lipids will be tested at baseline, 8th day and 3rd month, 6th month,12th month; hs-CRP will be tested at baseline and 8th day, 3rd month, Fg will be tested at baseline, 8th day, 3rd month. Safety will be also assessed by adverse event reports and clinical laboratory data including CK-MB, renal and hepatic function at 3rd month, 6th month,12th month.

Primary endpoint is the proportion of poor prognosis(modified Rankin scores>2) at 3 and 12 months post discharge. mRS scores>2 is defined as poor prognosis. And mRS scores≤2 scores were defined as good prognosis. Primary endpoint is the comparison of percentage of poor prognosis between two groups. Second endpoints include change from baseline in serum lipid, Fg and hs-CRP levels at 8th day, 3rd month, 6th month and 12th month after randomization. The incidence of vascular endpoint events including all-cause mortality, any event of recurrent ischemic stroke/TIA, hemorrhagic stroke, myocardial infarction and angina, and other noncerebral ischemia or hemorrhage. And change from admission in MMSE and Montreal scores of all subjects at 12th month.

Researchers who are responsible for evaluation of mRS, NIHSS scores, MMSE and Montreal scores will receive centralized training and be specialized. Specialized doctors follow-up the subjects with no knowledge of the statin therapies for the patients. Every month a meeting will be held to know if there are problems and to solve them.

Two special doctors in each center are responsible for follow-up visits. Patients will be asked to bring all empty packages to the clinic at each visit. The patient's compliance will be assessed by the investigator and recorded in the CRF. A pill count should be done at a patient level and recorded in the CRF and a dispensing log by the study site personnel.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Adults between 35 and 80 years old
3. Anterior circulation ischemic stroke within 72h of large arterial atherosclerosis subtype
4. First attack or without obvious sequelae after previous attacks of stroke(mRS≤1)
5. NIHSS score less than 24 when onset
6. Statin-naive(no statin therapy in the past 3 months)

Exclusion Criteria:

1. Familial hypercholesterolemia
2. Cardiogenic embolism and hemorrhagic transformation
3. Unknown cause and rare cause stroke subtypes
4. On or need to be on anticoagulant therapy
5. Severe hepatic(e.g. active liver disease, ALT or AST over 3 times of ULN), renal, hematopoietic, endocrine, myopathy , mental and cognitive diseases
6. Subjects with thrombolytic therapy
7. Concomitant treatment with ciclosporin
8. Allergy to statins or antiplatelet drugs
9. Planning to have a major operation or carotid ,vertebral angioplasty
10. Pregnancy and poor compliance.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with poor prognosis(modified Rankin scale>2) | 3rd month after onset of stroke
  A commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability, and it has become the most widely used clinical outcome measure for stroke clinical trials.mRS≤2 is defined as a good functional outcome, and mRS>2 is defined as a poor functional outcome.
proportion of patients with poor prognosis(modified Rankin scale>2) | 12th month after onset of stroke
  A commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability, and it has become the most widely used clinical outcome measure for stroke clinical trials.mRS≤2 is defined as a good functional outcome, and mRS>2 is defined as a poor functional outcome.

SECONDARY OUTCOMES:
the occurrence of vascular events( a composite) | 12th months after onset of stroke
  It includes all-cause mortality, any event of recurrent ischemic stroke/TIA, hemorrhagic stroke, myocardial infarction and angina, and other noncerebral ischemia or hemorrhage.
Change from baseline in cognitive function at 12 months | 12 months
  Mini-Mental State Examination and Montreal congnitive assessment

OTHER OUTCOMES:
Change from baseline in serum lipids(a composite) at 12 months | 3rd, 8th day and 3 rd, 6th and 12th month
  It includes cholesterol, low density lipoprotein and high density lipoprotein It includes cholesterol, triglycerides, high density lipoprotein, low density lipoprotein, hs-CRP and fibrinogen levels
Change from baseline in hs-CRP level at 3 months | baseline, 3rd, 6th and 12th month
  hs-CRP means hyper sensitive C-reactive protein
Change from baseline in Fg level at 3 months | 3rd month
  Fg means fibrinogen
Incidence of abnormal hepatic function(a composite) | 3rd month
  It includes elevation of hepatic enzymes(alanine aminotransferase and aspartate aminotransferase), jaundice, and hepatic failure.
Incidence of abnormal hepatic function(a composite) | 12th month
  It includes elevation of hepatic enzymes(alanine aminotransferase and aspartate aminotransferase), jaundice, and hepatic failure.
Incidence of renal dysfunction | 3rd month
  It includes elevation of serum creatinine levels and renal failure.
Incidence of renal dysfunction | 12th month
  It includes elevation of serum creatinine levels and renal failure.
Incidence of elevation of serum CK levels | 3rd month
  CK means creatine kinase
Incidence of elevation of serum CK levels | 12th month
  CK means creatine kinase

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Feng Liu, Ph.D,M.D., Study Chair — Second Afflilated Hospital of Soochow University
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

REFERENCES:
- [Background] Wang YJ, Zhang SM, Zhang L, Wang CX, Dong Q, Gao S, Huang RX, Huang YN, Lv CZ, Liu M, Qin HQ, Rao ML, Xiao Y, Xu YM, Yang ZH, Wang YJ, Wang CX, Wang JZ, Wang WZ, Wang J, Wang WJ, Wu J, Wu SP, Zeng JS, Zhang SM, Zhang L, Zhao XQ, Zhong LY. Chinese guidelines for the secondary prevention of ischemic stroke and transient ischemic attack 2010. CNS Neurosci Ther. 2012 Feb;18(2):93-101. doi: 10.1111/j.1755-5949.2011.00290.x. No abstract available. PMID 22313945
- [Background] Goldstein LB, Amarenco P, Zivin J, Messig M, Altafullah I, Callahan A, Hennerici M, MacLeod MJ, Sillesen H, Zweifler R, Michael K, Welch A; Stroke Prevention by Aggressive Reduction in Cholesterol Levels Investigators. Statin treatment and stroke outcome in the Stroke Prevention by Aggressive Reduction in Cholesterol Levels (SPARCL) trial. Stroke. 2009 Nov;40(11):3526-31. doi: 10.1161/STROKEAHA.109.557330. Epub 2009 Sep 10. PMID 19745172
- [Background] Kernan WN, Ovbiagele B, Black HR, Bravata DM, Chimowitz MI, Ezekowitz MD, Fang MC, Fisher M, Furie KL, Heck DV, Johnston SC, Kasner SE, Kittner SJ, Mitchell PH, Rich MW, Richardson D, Schwamm LH, Wilson JA; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Peripheral Vascular Disease. Guidelines for the prevention of stroke in patients with stroke and transient ischemic attack: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2014 Jul;45(7):2160-236. doi: 10.1161/STR.0000000000000024. Epub 2014 May 1. PMID 24788967
- [Background] Jauch EC, Saver JL, Adams HP Jr, Bruno A, Connors JJ, Demaerschalk BM, Khatri P, McMullan PW Jr, Qureshi AI, Rosenfield K, Scott PA, Summers DR, Wang DZ, Wintermark M, Yonas H; American Heart Association Stroke Council; Council on Cardiovascular Nursing; Council on Peripheral Vascular Disease; Council on Clinical Cardiology. Guidelines for the early management of patients with acute ischemic stroke: a guideline for healthcare professionals from the American Heart Association/American Stroke Association. Stroke. 2013 Mar;44(3):870-947. doi: 10.1161/STR.0b013e318284056a. Epub 2013 Jan 31. PMID 23370205
- [Background] Cimino M, Gelosa P, Gianella A, Nobili E, Tremoli E, Sironi L. Statins: multiple mechanisms of action in the ischemic brain. Neuroscientist. 2007 Jun;13(3):208-13. doi: 10.1177/1073858406297121. PMID 17519364
- [Background] Ni Chroinin D, Callaly EL, Duggan J, Merwick A, Hannon N, Sheehan O, Marnane M, Horgan G, Williams EB, Harris D, Kyne L, McCormack PM, Moroney J, Grant T, Williams D, Daly L, Kelly PJ. Association between acute statin therapy, survival, and improved functional outcome after ischemic stroke: the North Dublin Population Stroke Study. Stroke. 2011 Apr;42(4):1021-9. doi: 10.1161/STROKEAHA.110.596734. Epub 2011 Mar 3. PMID 21372311
- [Background] Calabro P, Yeh ET. The pleiotropic effects of statins. Curr Opin Cardiol. 2005 Nov;20(6):541-6. doi: 10.1097/01.hco.0000181482.99067.bf. PMID 16234628
- [Background] Ni Chroinin D, Asplund K, Asberg S, Callaly E, Cuadrado-Godia E, Diez-Tejedor E, Di Napoli M, Engelter ST, Furie KL, Giannopoulos S, Gotto AM Jr, Hannon N, Jonsson F, Kapral MK, Marti-Fabregas J, Martinez-Sanchez P, Milionis HJ, Montaner J, Muscari A, Pikija S, Probstfield J, Rost NS, Thrift AG, Vemmos K, Kelly PJ. Statin therapy and outcome after ischemic stroke: systematic review and meta-analysis of observational studies and randomized trials. Stroke. 2013 Feb;44(2):448-56. doi: 10.1161/STROKEAHA.112.668277. Epub 2013 Jan 3. PMID 23287777
- [Background] Blanco M, Nombela F, Castellanos M, Rodriguez-Yanez M, Garcia-Gil M, Leira R, Lizasoain I, Serena J, Vivancos J, Moro MA, Davalos A, Castillo J. Statin treatment withdrawal in ischemic stroke: a controlled randomized study. Neurology. 2007 Aug 28;69(9):904-10. doi: 10.1212/01.wnl.0000269789.09277.47. PMID 17724294
- [Background] Montaner J, Chacon P, Krupinski J, Rubio F, Millan M, Molina CA, Hereu P, Quintana M, Alvarez-Sabin J. Simvastatin in the acute phase of ischemic stroke: a safety and efficacy pilot trial. Eur J Neurol. 2008 Jan;15(1):82-90. doi: 10.1111/j.1468-1331.2007.02015.x. Epub 2007 Dec 7. PMID 18070096
- [Background] Sulter G, Steen C, De Keyser J. Use of the Barthel index and modified Rankin scale in acute stroke trials. Stroke. 1999 Aug;30(8):1538-41. doi: 10.1161/01.str.30.8.1538. PMID 10436097